CLINICAL TRIAL: NCT03327038
Title: Addressing Depression and Anxiety Symptoms in Patients With Inflammatory Bowel Disease (ADAPT-IBD)
Brief Title: Addressing Depression and Anxiety Symptoms in Patients With Inflammatory Bowel Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ADAPT-IBD
Record Dates: First submitted 2017-10-27; First posted 2017-10-31 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis; Depression; Anxiety
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychological Intervention (Experimental): Patients will be randomized to the intervention group after they have complete the study screening form. Patients randomized to the intervention group will receive a multifaceted intervention consisting of the following components (administered over an 8 week period): (1) Web-Based Cognitive Behavioral Therapy: (2) Short Questionnaires; (3) Ongoing Nurse Monitoring.
  Interventions: Behavioral: Web-Based Cognitive Behavioral Therapy; Other: Short Questionnaires; Behavioral: Nurse Monitoring; Other: Detailed Questionnaires; Other: Screening Form
- Control (Active Comparator): Patients will be randomized to the control group after they have completed the study screening form. Patients randomized to the control group will receive the usual standard of care that is available to patients with moderate anxiety or depression. Additionally, control patients will completed detailed questionnaires for assessment of primary and secondary outcomes.
  Interventions: Other: Detailed Questionnaires; Other: Screening Form

INTERVENTIONS:
Behavioral: Web-Based Cognitive Behavioral Therapy — Patients will receive access to a 5-week web-based CBT program entitled 'Mood Gym'. The program is derived from traditional, therapist-directed cognitive behavioral therapy. The program consists of 5 modules, and patients will asked to complete 1 module per week over, during weeks 2-6 over their intervention period.
  Arms: Psychological Intervention
Other: Short Questionnaires — Patients will receive emails to complete bi-weekly, web-based questionnaires at weeks 2, 4, and 6 of their intervention period. The short questionnaires will ask to patients to self-report their Depression (PHQ-9) and Anxiety (GAD-7) symptoms; along with their Crohn's Disease activity (PRO-2) or Ulcerative Colitis Disease Activity (MAYO-6).
  Arms: Psychological Intervention
Behavioral: Nurse Monitoring — Patient responses to the short questionnaires will be monitored by an IBD advanced practice nurse. The IBD nurse will determine if there are elevations in anxiety, depression, and disease activity over the intervention period. Based on patient responses to the short questionnaires, the nurse will follow-up with patients via email or telephone to address patient symptoms. If there are clinically important changes in the patients' disease activity the nurse may also arrange for the patients to receive expedited outpatient follow-up with their gastroenterologist.
  Arms: Psychological Intervention
Other: Detailed Questionnaires — Patients will complete a detailed questionnaires at enrollment (i.e. week 1 of enrollment) and also at post-intervention (i.e. week 8 of enrollment). The enrollment questionnaire will query the patients Ulcerative Colitis Disease Activity (MAYO-6) or Crohn's Disease Activity (PRO-2); Quality of Life (SIBDQ); and Patient Satisfaction with Health Care in IBD (CACHE). The post-intervention questionnaire will query the same information as the enrollment questionnaire but will also ask patients to self-report their depression (PHQ-9) and anxiety (GAD-7) symptoms.Quality of Life will be measured using the 10 item Short Inflammatory Bowel Disease Questionnaire (SIBDQ), which has a total score range of 10 to 70, with higher scores indicating better quality of life. Patient Satisfaction with Health Care in IBD will be measured using the 32 item CACHE Questionnaire, which scores from 0 -least satisfaction to 100-highest satisfaction.
Other: Screening Form — Patients will complete a screening form at routine IBD outpatient visits to Mount Sinai Hospital to self-report their depression and generalized anxiety symptoms. Their depression symptoms will be reported on the 9-item Patient Health Questionnaire (PHQ-9), which has a total score ranging from 0 to 27, with scores of 5, 10, 15 and 20 representing cut points for mild, moderate, moderately severe, and severe depression. Their generalized anxiety symptoms will be reported on the 7-item Generalized Anxiety Disorder Questionnaire (GAD-7), which has a total score ranging from 0 to 21, with scores of 5, 10, and 15 representing cut points for mild, moderate, and severe anxiety. Patients who self-report scores of moderate depression AND/OR moderate anxiety will be eligible to participate in this study.

SUMMARY:
Inflammatory Bowel Diseases (IBD) are chronic debilitating disorders of the gastrointestinal tract that comprise two subtypes; Crohn's Disease (CD) and Ulcerative Colitis (UC). Canada has among the highest incidence rates of CD and UC in the world, as high as 20.2 and 19.5 per 100,000 respectively. Although, IBD can occur at any age, it is frequently diagnosed in the second and third decades of life, at a time when vulnerable individuals are entering the prime years of their lives. This age of onset, coupled with the recurrent and frequently relapsing nature of these disorders, can significantly impair the psychological well-being of patients. Therefore, it's not surprising that patients with IBD report a higher burden of depression and anxiety in comparison to the general population. The prevalence of depression and anxiety in patients with IBD have previously been linked to the following: (1) Increased risk of surgery; (2) Increased number of relapses; (3) Clinical recurrence; (4) Treatment failure and earlier retreatment; (5) Lower self-reported quality of life, satisfaction, and medication adherence; (6) and Increased health care utilization. Although, depression and anxiety are highly treatable conditions, they are often under-recognized and under- treated in patients with IBD. The most common treatments for these disorders are pharmacological agents and psychological treatments. Psychological treatments like Cognitive Behavioral Therapy (CBT) have extensive support for treatment of depression and anxiety. The major advantage of psychological treatments over pharmacological agents is their ability to sustain improved depression and anxiety symptoms in patients post-treatment. As part of this study, we aim to evaluate the following:

Specific Aim #1: Determine whether a psychological intervention, involving web-based CBT, is effective in ameliorating depression and anxiety symptoms in a cohort of adult IBD patients.

Specific Aim #2: Determine the durability effect of the intervention on sustaining improved psychiatric symptoms.

Specific Aim #3: Determine the impact of a psychological on IBD-specific and psychiatric-specific health care utilization.

DETAILED DESCRIPTION:
Inflammatory Bowel Diseases (IBD) are chronic debilitating disorders of the gastrointestinal tract that comprise two subtypes; Crohn's Disease (CD) and Ulcerative Colitis (UC). Canada has among the highest incidence rates of CD and UC in the world, as high as 20.2 and 19.5 per 100,000 respectively. Although, IBD can occur at any age, it is frequently diagnosed in the second and third decades of life; at a time when vulnerable individuals are entering the prime years of their lives. This age of onset, coupled with the recurrent and frequently relapsing nature of these disorders, can significantly impair the psychological well-being of patients. Therefore, it's not surprising that patients with IBD report a higher burden of depression and anxiety in comparison to the general population.

The rates of depression in patients with IBD, as measured by the National Population Health Survey and the Canadian Community Health Survey, range from 14.7% to 16.3%. These rates are significantly higher than the general Canadian population, in which 5.6% of healthy respondents reported a 12-month prevalence of depression. Moreover, studies among clinical samples of IBD patients have reported rates of depression as high as 35%. The prevalence of depression and anxiety in patients with IBD have previously been linked to the following: (1) Increased risk of surgery; (2) Increased number of relapses; (3) Clinical recurrence; (4) Treatment failure and earlier retreatment; (5) Lower self-reported quality of life, satisfaction, and medication adherence; (6) and Increased health care utilization.

Although, depression and anxiety are highly treatable conditions, they are often under recognized and under treated in patients with IBD. The most common treatments for these disorders are pharmacological agents and psychological treatments. Psychological treatments like Cognitive Behavioral Therapy (CBT) have extensive support for treatment of depression and anxiety. CBT refers to a group of interventions that share the notion that cognitive factors influence mental disorders and psychological distress, and that maladaptive cognitions contribute to emotional distress and behavioral problems. The major advantage of psychological treatments over pharmacological agents is their ability to sustain improved depression and anxiety symptoms in patients post-treatment.

Considering the prevalence and impact of depression and anxiety disorders in patients with IBD, further research in this area is needed to identify the most effective approaches for screening and treatment of these disorders. Research is also need to ascertain the effects of psychological treatments for depression and anxiety on influencing physiological aspects of IBD. As part of this study, we aim to evaluate the effectiveness of a psychological intervention which incorporates web-based CBT intervention on a cohort of adult IBD patients; by measuring its impact on clinical and self-reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* PHQ-9 AND/OR GAD-7 score ≥ 10
* Confirmed diagnosis of IBD (based on record of diagnostic endoscopy)
* Access to Computer or Smartphone
* Access to an Internet Connection

Exclusion Criteria:

* Patients without a record of diagnostic endoscopy in their clinical record
* Under psychological treatment parallel to the intervention being carried out
* Diagnosis of major depressive, dysthymic, bipolar or psychotic disorder
* History of anti-depressant medication use within 1 month of enrollment
* History of substance abuse or dependence within 1 month of enrollment
* Previous course of CBT within 12 months of Enrollment
* History of suicide
* History of psychiatric hospitalization
* Inability to provide informed consent
* Insufficient command of written and spoken English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-05-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Rates of Moderate Depression (PHQ-9) | Post-Intervention (i.e. week 8)
  Post-intervention rates will be compared between study groups
Rates of Moderate Anxiety (GAD-7) | Post-Intervention (i.e. week 8)
  Post-intervention rates will be compared between study groups
Rates of Moderate Depression (PHQ-9) and co-morbid Anxiety (GAD-7) | Post-Intervention (i.e. week 8)
  Post-intervention rates will be compared between study groups

SECONDARY OUTCOMES:
Difference in Depression Scores (PHQ-9) | Post-Intervention (i.e. week 8)
  Post-intervention Patient Health Questionnaire (PHQ-9) scores will be compared between study groups
Difference in Anxiety Scores (GAD-7) | Post-Intervention (i.e. week 8)
  Post-intervention Generalized Anxiety Disorder (GAD-7) scores will be compared between study groups
Change in Depression Scores (PHQ-9) | Between Enrollment (i.e. week 1) and Post-intervention (i.e. week 8)
  Change in Patient Health Questionnaire (PHQ-9) scores between enrollment and post-intervention will be compared within study groups
Change in Anxiety Scores (GAD-7) | Between Enrollment (i.e. week 1) and Post-intervention (i.e. week 8)
  Change in Generalized Anxiety Disorder (GAD-7) scores between enrollment and post-intervention will be compared within study groups
Rates of Active IBD (PRO-2 or MAYO-6) | Post-Intervention (i.e. week 8)
  Post-intervention rates will be compared between study groups
Rates of Active IBD (PRO-2 or MAYO-6) | Between Enrollment (i.e. week 1) and Post-intervention (i.e. week 8)
  Change in rates between enrollment and post-intervention will be compared within study groups
Difference in Quality of Life Scores (SIBDQ) | Post-Intervention (i.e. week 8)
  Post-intervention Short Inflammatory Bowel Disease Questionnaire (SIBDQ) scores will be compared between study groups
Difference in Patient Satisfaction Scores (CACHE) | Post-Intervention (i.e. week 8)
  Post-intervention Patient Satisfaction with Health Care in IBD (CACHE) scores will be compared between study groups
Change in Quality of Life Scores (SIBDQ) | Between Enrollment (i.e. week 1) and Post-intervention (i.e. week 8)
  Change in Short Inflammatory Bowel Disease Questionnaire (SIBDQ) scores between enrollment and post-intervention will be compared within study groups
Change in Patient Satisfaction Scores (CACHE) | Between Enrollment (i.e. week 1) and Post-intervention (i.e. week 8)
  Change in Patient Satisfaction with Health Care in IBD (CACHE) scores between enrollment and post-intervention will be compared within study groups
Rates of IBD-related hospitalizations | Between Enrollment (i.e. week 1) and Post-intervention (i.e. week 8)
  Event rates over trial period will be compared between study groups
Rates of IBD-related surgery over intervention period | Between Enrollment (i.e. week 1) and Post-intervention (i.e. week 8)
  Event rates over trial period will be compared between study groups

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey C Nguyen, MD, PhD, Principal Investigator — Mount Sinai Hospital (Toronto, ON, Canada)
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Yanartas O, Kani HT, Bicakci E, Kilic I, Banzragch M, Acikel C, Atug O, Kuscu K, Imeryuz N, Akin H. The effects of psychiatric treatment on depression, anxiety, quality of life, and sexual dysfunction in patients with inflammatory bowel disease. Neuropsychiatr Dis Treat. 2016 Mar 24;12:673-83. doi: 10.2147/NDT.S106039. eCollection 2016. PMID 27069364
- [Background] Bernstein CN, Wajda A, Svenson LW, MacKenzie A, Koehoorn M, Jackson M, Fedorak R, Israel D, Blanchard JF. The epidemiology of inflammatory bowel disease in Canada: a population-based study. Am J Gastroenterol. 2006 Jul;101(7):1559-68. doi: 10.1111/j.1572-0241.2006.00603.x. PMID 16863561
- [Background] Graff LA, Walker JR, Bernstein CN. Depression and anxiety in inflammatory bowel disease: a review of comorbidity and management. Inflamm Bowel Dis. 2009 Jul;15(7):1105-18. doi: 10.1002/ibd.20873. PMID 19161177
- [Background] Sajadinejad MS, Asgari K, Molavi H, Kalantari M, Adibi P. Psychological issues in inflammatory bowel disease: an overview. Gastroenterol Res Pract. 2012;2012:106502. doi: 10.1155/2012/106502. Epub 2012 Jun 21. PMID 22778720
- [Background] Fiest KM, Walker JR, Bernstein CN, Graff LA, Zarychanski R, Abou-Setta AM, Patten SB, Sareen J, Bolton JM, Marriott JJ, Fisk JD, Singer A, Marrie RA; CIHR Team Defining the Burden and Managing the Effects of Psychiatric Comorbidity in Chronic Immunoinflammatory Disease. Systematic review and meta-analysis of interventions for depression and anxiety in persons with multiple sclerosis. Mult Scler Relat Disord. 2016 Jan;5:12-26. doi: 10.1016/j.msard.2015.10.004. Epub 2015 Oct 19. PMID 26856938
- [Background] Fuller-Thomson E, Sulman J. Depression and inflammatory bowel disease: findings from two nationally representative Canadian surveys. Inflamm Bowel Dis. 2006 Aug;12(8):697-707. doi: 10.1097/00054725-200608000-00005. PMID 16917224
- [Background] Hofmann SG, Asnaani A, Vonk IJ, Sawyer AT, Fang A. The Efficacy of Cognitive Behavioral Therapy: A Review of Meta-analyses. Cognit Ther Res. 2012 Oct 1;36(5):427-440. doi: 10.1007/s10608-012-9476-1. Epub 2012 Jul 31. PMID 23459093
- [Background] Szigethy E, Kenney E, Carpenter J, Hardy DM, Fairclough D, Bousvaros A, Keljo D, Weisz J, Beardslee WR, Noll R, DeMASO DR. Cognitive-behavioral therapy for adolescents with inflammatory bowel disease and subsyndromal depression. J Am Acad Child Adolesc Psychiatry. 2007 Oct;46(10):1290-1298. doi: 10.1097/chi.0b013e3180f6341f. PMID 17885570
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391